CLINICAL TRIAL: NCT02587624
Title: Safety, Radiation Exposure and Efficacy of Remote MAGNetic Catheter Ablation for Atrial Fibrillation
Brief Title: Remote MAGNetic Catheter Ablation for Atrial Fibrillation
Acronym: MAGNA-AF
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Dr. Dirk Bastian, Principle investigator, Paracelsus Medical University
Other Study IDs: PMUN-DB-002-MAGNA-AF
Record Dates: First submitted 2015-10-18; First posted 2015-10-27 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; remote magnetic navigation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RMN AF ablation: Consecutive patients with class I or class IIa indication for catheter ablation for symptomatic atrial fibrillation according to the current guidelines.
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — Intervention: All patients undergo magnetically guided pulmonary vein antral isolation and mapping for fibrotic areas. Procedural endpoint: bidirectional PV block. Additional substrate modification on decision of the operator.

SUMMARY:
Prospective observational single center trial, evaluating the safety, radiation exposure and efficacy of remote magnetic catheter ablation for atrial fibrillation in daily routine.

DETAILED DESCRIPTION:
Background: Since the first description in 1998 catheter-interventional ablation (CA) has evolved to a standard treatment for symptomatic drug-refractory atrial fibrillation (AF).

Ablation efficacy but also complication percentage and radiation exposure are influenced by several factors, among them patient age, body weight, type and duration of AF, underling cardiac disease as well as the used ablation method, technology and the experience of the operator.

The objectives of developing a system for remote magnetic catheter navigation (RMN) were to improve the efficacy and safety of complex ablation procedures and to reduce radiation exposure. However, convincing data supporting this theory are still lacking.

Aim: To evaluate efficacy, safety profile / complication rate and radiation exposure in serial ablation procedures for paroxysmal and persistent AF as well as repeat interventions based on remote magnetic navigation and 3-D image integration with assessment of the learning curve for this complex technology.

Design: single center observational registry, analytical questioning, non-randomized, non-controlled, not blinded, consecutive patient inclusion

Study population:

Inclusion criteria: Consecutive patients with class I or class IIa indication for CA for symptomatic atrial fibrillation according to the current guidelines.

Exclusion criteria:

* Contraindication for AF catheter ablation
* Contraindication for RMN procedure. (These patients may undergo AF ablation with another technology, e.g. cryo-balloon ablation).
* Age < 18 years, gravidity

Endpoints Primary endpoint

Safety:

* The number of peri-procedural major complications.
* Adverse events are classified according to the 2012 Expert consensus statement on catheter and surgical ablation of AF [Calkins H et al. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation. Europace (2012) 14, 528-606 doi:10.1093/europace/eus027].

Secondary endpoints Efficacy

* Acute: number of successfully isolated pulmonary veins.
* Mid-term: freedom from any atrial tachyarrhythmia (atrial fibrillation/atypical atrial flutter/atrial tachycardia; duration > 30 sec) after 6 months follow-up (initial blanking period of 3 months).
* Long-term:
* Freedom from any atrial tachyarrhythmia (duration > 30 sec) after 12 months follow-up (initial blanking period of 3 months).
* Time to first recurrence of an atrial tachyarrhythmia after an initial blanking period of 3 months.

Radiation exposure:

* mean effective dose (ED), based on the measured dose-area-product. Aim is to show the potential of RMN to reduce the mean ED below 1.5 mSv in daily routine RMN AF ablation procedures
* The fluoroscopy parameters are documented for system calibration (A), transseptal access/catheter positioning (B), mapping/ablation (C).

Safety:

* Number of peri-procedural minor complications
* Number of all procedure-related complications during 12 months follow-up.

Subgroups:

* Type of AF (paroxysmal versus non-paroxysmal)
* Type of antiarrhythmic drug treatment (AAD)
* Demonstration of low-voltage areas / fibrosis
* Ablation: only pulmonary vein antral isolation (PVAI) versus additional substrate modification / box isolation of fibrotic areas (BIFA)
* Adipositas (BMI ≥ 30 kg/m²)
* Transseptal access after puncture versus via patent foramen ovale
* First ablation versus repeat procedure

Randomisation: none

Study procedure:

Pre-ablation: screening of all patients, referred for catheter ablation for AF. Inclusion after given informed consent. Oral anticoagulation (OAC) for at least 3 weeks. Transesophageal echocardiography (TEE) in all patients.

Ablation: Non-interrupted OAC, non-vitamin-K antagonist treatment withheld only the morning before ablation. All patients undergo PVAI and mapping for fibrotic areas, additional substrate modification on decision of the operator.

Techniques and technologies used: RMN: Niobe/Epoch®, Navigant™, 0.1 Tesla, Stereotaxis Inc.; fluoroscopy system: Siemens AXIOM-Artis VC12B, 6-1 fps; non-fluoroscopic mapping (NFM): Carto-RMT, magnetic resonance-image-integration, (Biosense-Webster Inc.); TEE-guided single transseptal puncture, "Single catheter ablation" technique: Navistar-RMT Thermocool (Biosense-Webster Inc.), target temperature 48°C, power limit 40Watts (posterior left atrial wall) up to 50W, irrigation infusion rate 17 mL/min; Heparin for maintaining an activated clotting time between 300 to 400 sec. Endpoint: bidirectional PV-block.

Post-ablation in hospital: OAC continued immediately following sheath removal after ablation for a minimum of 2 months, thereafter according to embolic risk (CHA2DS2-VASc-risk evaluation). 48 hours telemonitoring, echocardiography.

Follow up: blanking period 3 months. Clinical evaluation after 3, 6 and 12 months including echocardiography and 72-hours Holter.

Unscheduled visits for complications and symptoms suggesting recurrent tachyarrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with class I or class IIa indication for catheter ablation for symptomatic atrial fibrillation according to the current guidelines.

Exclusion Criteria:

* Contraindication for AF catheter ablation
* Contraindication for magnetically guided ablation procedure
* Age < 18 years, gravidity, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with class I or class IIa indication for catheter ablation for symptomatic atrial fibrillation according to the current guidelines [Camm AJ et al. 2012 focused update of the ESC guidelines for the management of atrial fibrillation. European Heart Journal (2012) 33, 2719-2747].
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2011-03; Primary Completion 2025-09 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Safety: peri-procedural major complications. | Peri-procedural (from the beginning of the procedure until 48 hours after sheath removal)
  Procedure associated adverse events are classified according to the 2012 Expert consensus statement on catheter and surgical ablation of AF [Calkins et al, Europace 2012].

SECONDARY OUTCOMES:
Acute efficacy: number of successfully isolated pulmonary veins. | Intra-procedural
  Number of successfully isolated pulmonary veins.
Long-term efficacy: freedom from atrial tachyarrhythmia. | 12 months
  - Freedom from any atrial tachyarrhythmia (AF/flutter/atrial tachycardia; duration > 30 sec, initial blanking period of 3 months).
Long-term efficacy: time to recurrence of atrial tachyarrhythmia. | 12 months
  - Time to first recurrence of any atrial tachyarrhythmia (AF/flutter/atrial tachycardia; duration > 30 sec) after an initial blanking period of 3 months
Safety: radiation exposure. | Peri-procedural (from the beginning of the procedure until sheath removal)
  * mean effective dose (ED), based on the measured dose-area-product. Aim is to show the potential of RMN to reduce the mean ED below 1.5 mSv in daily routine RMN AF ablation procedures
  * The fluoroscopy parameters are documented for system calibration (A), transseptal access/catheter positioning (B), mapping/ablation (C).
Safety: peri-procedural minor complications. | Peri-procedural (from the beginning of the procedure until 48 hours after sheath removal)
  Procedure related adverse events are classified according to the 2012 Expert consensus statement on catheter and surgical ablation of AF [Calkins et al, Europace 2012].
Safety: incidence of procedure related adverse events during long term follow-up. | 12 months
  Any complication during follow-up. Procedure related adverse events are classified according to the 2012 Expert consensus statement on catheter and surgical ablation of AF [Calkins et al, Europace 2012].

OTHER OUTCOMES:
Efficacy: freedom from atrial tachyarrhythmia in pre-specified patient subgroups. | 12 months
  Freedom from any atrial tachyarrhythmia (AF/flutter/atrial tachycardia; duration > 30 sec, initial blanking period of 3 months) in different subgroups:
  * Type of AF (paroxysmal versus non-paroxysmal)
  * Type of antiarrhythmic drug treatment
  * Demonstration of low-voltage areas / fibrosis
  * Ablation: only pulmonary vein antral isolation (PVAI) versus additional substrate modification / box isolation of fibrotic areas (BIFA)
  * Adipositas (BMI ≥ 30 kg/m²)
  * Transseptal access after puncture versus via patent foramen ovale
  * First ablation versus repeat procedure
Efficacy: time to first recurrence of atrial tachyarrhythmia in pre-specified patient subgroups. | 12 months
  Time to first recurrence of any atrial tachyarrhythmia (AF/flutter/atrial tachycardia; duration > 30 sec) after an initial blanking period of 3 months in different subgroups:
  * Type of AF (paroxysmal versus non-paroxysmal)
  * Type of antiarrhythmic drug treatment
  * Demonstration of low-voltage areas / fibrosis
  * Ablation: only pulmonary vein antral isolation (PVAI) versus additional substrate modification / box isolation of fibrotic areas (BIFA)
  * Adipositas (BMI ≥ 30 kg/m²)
  * Transseptal access after puncture versus via patent foramen ovale
  * First ablation versus repeat procedure
Safety: procedure related complications in pre-specified subgroups during long term follow-up. | 12 months
  Number of procedure associated complications in different subgroups:
  * Type of AF (paroxysmal versus non-paroxysmal)
  * Type of antiarrhythmic drug treatment
  * Demonstration of low-voltage areas / fibrosis
  * Ablation: only pulmonary vein antral isolation (PVAI) versus additional substrate modification / box isolation of fibrotic areas (BIFA)
  * Adipositas (BMI ≥ 30 kg/m²)
  * Transseptal access after puncture versus via patent foramen ovale
  * First ablation versus repeat procedure
Radiation exposure in pre-specified patient subgroups. | Intra-procedural (duration of procedure)
  Procedural radiation exposure in different subgroups:
  * Type of AF (paroxysmal versus non-paroxysmal)
  * Demonstration of low-voltage areas / fibrosis
  * Ablation: only pulmonary vein antral isolation (PVAI) versus additional substrate modification / box isolation of fibrotic areas (BIFA)
  * Adipositas (BMI ≥ 30 kg/m²)
  * Transseptal access after puncture versus via patent foramen ovale
  * First ablation versus repeat procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bastian, MD, Study Chair — Klinikum Fuerth, Fuerth
Locations (1):
- Paracelsus Medical University, Klinikum Nürnberg, Nuremberg, Bavaria, Germany

REFERENCES:
- [Background] Bastian D, Schwab J, Steurer KT, Brinker-Paschke A, Boessenecker A, Doering R, Karakurt Z, Vitali-Serdoz L, Pauschinger M, Gohl K. Oesophageal injury following magnetically guided single-catheter ablation for atrial fibrillation: insights from the MAGNA-AF registry. Europace. 2018 May 1;20(suppl_2):ii48-ii55. doi: 10.1093/europace/euy021. PMID 29722860